CLINICAL TRIAL: NCT05466175
Title: A Multicenter, Prospective Clinical Study of Olverembatinib Combined With Chemotherapy in the Treatment of de Novo Adult Philadelphia Chromosome-positive Acute Lymphoid Leukemia
Brief Title: A Study of Olverembatinib in the Treatment of Ph+ ALL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chen Suning (Other)
Responsible Party: Sponsor-Investigator, Chen Suning, Physician, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ-ALL01
Record Dates: First submitted 2022-07-04; First posted 2022-07-20 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-07

CONDITIONS: Philadelphia-Positive ALL
Keywords: Olverembatinib, Ph+ALL, adult, de novo
MeSH Terms: interventions — olverembatinib; Prednisone; Vincristine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): combination of Olverembatinib with chemotherapy
  Interventions: Drug: Olverembatinib; Drug: Prednisone; Drug: Vincristine

INTERVENTIONS:
Drug: Olverembatinib — Given PO
Drug: Prednisone — Given Intravenous
Drug: Vincristine — Given Intravenous

SUMMARY:
In this study, adults with newly-diagnosed Philadelphia Chromosome-positive acute lymphoblastic leukemia (Ph+ ALL) will receive first-line therapy of a novel third-generation TKI Olverembatinib.

The main purpose of the study is to evaluate the efficacy and safety of Olverembatinib in Ph+ ALL patients.

DETAILED DESCRIPTION:
Eligible participants will receive an 28-day induction regimen of Olverembatinib (40mg, QOD) combined with VP-chemotherapy, followed by 4 cycles of Hyper-CVAD A/B treatment (each lasting 28 days). If complete molecular response (CMR) is achieved at the 3rd month, participants will receive another three cycles of Hyper-CVAD A/B treatment. Maintenance therapy would be given for at least 1 year with monthly courses of vincristine, prednisone and Olverembatinib. If participants fail to achieve CMR at the 3rd month, or patients with an available matched donor had the option to proceed to allogeneic stem cell transplantation (allo-HSCT) at the discretion of the treating physician. Olverembatinib would be administered at the time of hematopoietic reconstruction for at least 1 year.

Intrathecal injection would be performed on day 15 of induction therapy and before each course of consolidation therapy to prevent central nervous system leukemia (CNSL).

It is expected that about 55 patients will take part in this study.

ELIGIBILITY:
Inclusion Criteria

1. Male or non-pregnant, non-lactating female patients who are 18 years of age or older.
2. Newly diagnosed Philadelphia chromosome-positive (Ph+) or BCR-ABL1-positive ALL, as defined by the 2016-WHO criteria. Participants should not be treated with any kind of TKIs or chemotherapy. Participants who only received preconditioning can be enrolled.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, and expected survival period ≥ 3 months.
4. Organ function as indicated by the following laboratory indicators must be met:

1) Alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) ≤ 2.5 × ULN; 2) Total bilirubin≤1.5×ULN; 3) Serum creatinine≤1.5×ULN or 24-hour calculated creatinine clearance≥50mL/min when serum creatinine >1.5×ULN; 4) Amylase≤1.5×ULN, lipase≤1.5×ULN; 5) Cardiac ejection fraction (EF) > 50%, pulmonary artery systolic blood pressure ≤ 50mmHg; 6) QT interval corrected on electrocardiogram (ECG) evaluation: QTc≤450ms in males or ≤470ms in females; 7) PT, APTT and INR≤1.5×ULN.

5. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. The presence of central nervous system (CNS) or testicular active ALL.
2. Human immunodeficiency virus (HIV) infection, or chronic infection with hepatitis B virus (HBsAg positive) or hepatitis C virus (anti-HCV positive).
3. Uncontrolled active infection.
4. Patients who are currently suffering from active autoimmune disease or a history of autoimmune disease potentially involving the CNS.
5. Patients who have a history of clinically significant CNS lesions or is currently suffering from clinically significant CNS lesions.
6. Patients who have any history of heart or vascular disease, such as hypertension (systolic blood pressure(HBP) > 140mmHg and/or diastolic blood pressure > 90mmHg), or take medications that are known to cause QT interval prolongation. The patients with well controlled HBP can be considered to be included.
7. Cardiac ultrasonography indicates that pulmonary artery systolic blood pressure is >50 mmHg; or there are clinical symptoms related to pulmonary arterial hypertension.
8. Patients who suffer from severe bleeding disorders unrelated to Ph+ ALL.
9. Patients who have any other malignant tumors that require treatment.
10. Patients who have a history of pancreatitis or a history of alcohol abuse.
11. Patients who have severe hypertriglyceridemia (triglyceride ≥ 5.6mmol/L).
12. Patients who are pregnant, planning to become pregnant or breastfeeding.
13. Patients who underwent major surgery (except for minor surgery such as catheter placement or bone marrow biopsy) within 14 days before the first drug.
14. Patients who may not be able to complete all study visits or procedures required by the study protocol, including follow-up visits, and/or fail to comply with all required study procedures.
15. Patients who suffer from any condition or illness that, in the opinion of the Investigator, would compromise patient safety or interfere with the evaluation of the safety of the research drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Complete Molecular Remission | From Induction through the end of one cycle of Hyper-CVAD A and B (approximately 3 months) (Cycle length is equal to [=] 28 days) ]
  Will be estimated along with the 95% credible intervals.

SECONDARY OUTCOMES:
Percentage of Participants with CR and Incomplete Complete Remission (CRi) | At the end of consolidation therapy (approximately 9 months) and one year after allo-HSCT
  Will be estimated along with the 95% credible intervals.
Duration of Complete Molecular Remission | From the date of acquisition of complete molecular remission until the date of loss of complete molecular remission, assessed up to 2 to 4 years.
  Will be estimated along with the 95% credible intervals.
Event-free survival (EFS) | From the first day of treatment until any failure (resistant disease, relapse, or death), assessed up to 2 to 4 years ]
  The Kaplan-Meier method will be used to assess EFS probabilities.
Overall survival (OS) | From the first day of treatment to time of death from any cause, assessed up 2 to 4 years.
  The Kaplan-Meier method will be used to assess OS probabilities.
Incidence of adverse events (AEs) | Up to approximately 2 to 4 years
  Will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The proportion of patients with AEs will be estimated, along with the Bayesian 95% credible interval.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China